CLINICAL TRIAL: NCT05669027
Title: Effective Self-Management of Chronic Pain With mHealth Neurofeedback
Brief Title: Mobile Neurofeedback for Low Back Pain
Acronym: NINR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00108939; 1R01NR019788-01A1 (NIH)
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low Back Pain
Keywords: Neurofeedback; Biofeedback; Mobile Device; chronic low back pain; Pain Intensity; Relaxation; mHealth; Opioid
MeSH Terms: conditions — Pain | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: Examine effects of mobile neurofeedback on changes in pain intensity, pain interference, physical function, and EEG alpha (8-13 Hz) power.
  Examine mediating effect of self-efficacy on changes in pain outcomes.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental Condition (Experimental): Mobile Neurofeedback intervention arm
  Interventions: Device: Neurofeedback
- Control Condition (Placebo Comparator): Sham-control arm
  Interventions: Device: Sham (Placebo Control)

INTERVENTIONS:
Device: Neurofeedback — Participants will be asked to complete 10-minute sessions at least 4 days per week for 12 weeks. Participants will be asked to report their current level of pain, stress, and anger before and after each session. The experimental condition involves a mobile app that provides auditory feedback signaling EEG alpha power above a threshold level, denoting a physiologically relaxed state.
  Arms: Experimental Condition
Device: Sham (Placebo Control) — Participants will be asked to complete 10-minute sessions at least 4 days per week for 12 weeks. Participants will be asked to report their current level of pain, stress, and anger before and after each session. The control condition involves a visually identical mobile app yoked to a pre-recorded set of actual neurofeedback sessions (i.e., placebo).
  Arms: Control Condition

SUMMARY:
The purpose of this study is to learn more about improving the quality of treatments for people who have chronic low back pain. Participants will complete interviews with Duke researchers at four different time points: the beginning of the study, at 3 months, at 6 months, and at 9 months. Participants will be asked to use a mobile app and a headset that are designed to train the brain to be more relaxed. Participants will use the mobile app for 10 minutes at a time, four times a week for three months. The study team will also check in with participants about app use six times throughout the study, via phone or video conference.

DETAILED DESCRIPTION:
This is a double-blind randomized controlled trial to test effects of mHealth mobile neurofeedback on the outcomes of pain, enrolling 150 adult participants (18 years of age or older) with chronic low backpain. Participants will be scheduled for a baseline interview at Dr. Elbogen's research office at Duke after a preliminary telephone screen. After providing informed consent, participants will complete an eligibility assessment, a physical function test, self-report questionnaire on pain interference including clinical interviews for health outcomes of pain; self-report questionnaire on pain interference, pain self-efficacy, drug and alcohol use, opioid use, drug/alcohol use; a physical function test; and an EEG. Participants will be be randomly assigned to either an experimental (mobile neurofeedback) or placebo-control (sham neurofeedback) group. All participants will receive a portable Muse EEG headset and an iPod Touch with a mobile app named 'Mobile Neurofeedback' and be asked to complete 10-minute sessions at least 4 days per week for 12 weeks. Participants will be asked to report their current level of pain, stress, and anger before and after each session. The experimental condition involves a mobile app that provides auditory feedback signaling EEG alpha power above a threshold level, denoting a physiologically relaxed state. The control condition involves a visually identical mobile app yoked to a pre-recorded set of actual neurofeedback sessions (i.e., placebo). Study coordinators will conduct 6 check in calls in the intervening period, the study team will to reinforce training, troubleshoot technical problems, and assess any risk/safety issues (weeks 1,3,5,7,9, and 11). Follow-up data will be collected upon completion of the intervention at 12 weeks, 24 weeks and 36 weeks. During all follow-up visits, participants will complete self-report questionnaires, a physical function test, and an EEG. Data will be collected at baseline, 3, 6, and 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. Responding greater than 3 months to "How long has low back pain been an ongoing problem for you?"
2. Responding 'at least half the days' to "How often has low back pain been an ongoing problem for you over the past 6 months?"

Investigators will follow recommendations to items and responses provided by the NIH Task Force on Research Standards for Chronic Low Back Pain, which specifically: "recommended 2 questions to achieve the definition of chronic low back pain: (1) How long has back pain been an ongoing problem for you? (2) How often has low back pain been an ongoing problem for you over the past 6 months? A response of greater than 3 months to question 1 and a response of 'at least half the days in the past 6 months' to question 2 would define chronic lower back pain."

Exclusion Criteria:

1. History of seizures.
2. Planning pain-related surgery in the next 9 months.
3. Individuals with implanted medical devices that could experience interference during EEG and/or ECG, such as a spinal cord stimulator or pacemaker.
4. Lower back pain is associated with compensation or litigation issues.
5. Rating of past week pain intensity<4 on 0-10 point scale.
6. Rating of past week pain interference<4 on 0-10 point scale.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | Months 3, 6, and 9
  Low back pain intensity on a 0-10 point rating scale, where higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Change in pain interference as measured by PROMIS (Patient-Reported Outcomes Measurement Information System) | Months 3, 6, and 9
  A higher PROMIS T-score indicates greater pain interference. The minimum score is 8 and the maximum score is 40.
Change in physical function as measured by speed on the 50-foot walk test | Months 3, 6, and 9
  Participant is timed by how long it takes for them to walk 50 feet.
Change in alpha brainwave (8 - 13 Hz) power as measured by EEG (electroencephalography) | Months 3, 6, and 9
  An EEG can identify and measure the electrical activity in the brain. Higher EEG alpha brainwave power indicates a greater state of relaxation.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Elbogen, Ph.D., Principal Investigator — Duke - Professor in Psychiatry and Behavioral Sciences
Locations (1):
- Duke University Medical Center, Department of Psychiatry, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No